CLINICAL TRIAL: NCT00027898
Title: A Phase I Study of PS-341 (NSC 681239), Carboplatin, and Etoposide in Patients With Advanced Solid Tumors Refractory to Standard Therapy
Brief Title: Bortezomib and Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02432; COMIRB 01-288; U01CA099176 (NIH); CDR0000069091 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Bortezomib; Carboplatin; Etoposide

ARMS (1):
- Treatment (bortezomib, carboplatin, and etoposide) (Experimental): Patients receive bortezomib IV on days 1 and 8, carboplatin IV over 30 minutes on day 1, and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Drug: carboplatin; Drug: etoposide; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Phase I trial to study the effectiveness of combining bortezomib with carboplatin and etoposide in treating patients who have advanced solid tumors that have not responded to previous treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of bortezomib, carboplatin, and etoposide in patients with advanced solid tumors refractory to standard therapy.

II. Evaluate biologic effects of bortezomib on relevant targets in the tumor tissues of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of bortezomib, etoposide, and carboplatin.

Patients receive bortezomib IV on days 1 and 8, carboplatin IV over 30 minutes on day 1, and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 6 additional patients with newly diagnosed, chemotherapy-naive extensive stage small cell lung cancer, and 6 patients with other tumor types, are treated at that dose.

PROJECTED ACCRUAL: A total of 12-27 patients will be accrued for this study within 6-14 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor cancer for which no curativetherapy exists
* Clinically stable CNS disease is allowed provided the following criteria are met:

  * No uncontrolled brain metastases or CNS involvement
  * No active seizures
  * On stable dose of antiseizure or steroid medication for at least 7 days before study enrollment
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 9 g/dL
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No other serious concurrent systemic disorders (including other malignancy)
* No prior bone marrow or peripheral blood stem cell transplantation
* No concurrent immunotherapy
* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior carboplatin and/or etoposide allowed
* No more than 2 prior courses of mitomycin
* See Disease Characteristics
* No concurrent hormonal therapy
* At least 4 weeks since prior radiotherapy and recovered
* Palliative radiotherapy involving less than 35% bone marrow reserve allowed if completed at least 2 weeks before study enrollment
* No prior wide-field radiotherapy to 35% or more of bone marrow
* No prior pelvic radiotherapy
* No concurrent radiotherapy
* At least 28 days since prior investigational agents
* No other concurrent experimental medications

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-01; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level below the dose level that results in DLT in >= 2 of 6 new patients assessed using NCI CTC version 2.0 | 21 days
Biological data | Up to 4 years
  The variation of these samples as a function of dose and time will be analyzed to define the mathematical function (e.g. linear, exponential, logistic) that best fits and models the data.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Gore, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States